CLINICAL TRIAL: NCT00995878
Title: The FIRSTT Study: Comparing Focused Ultrasound and Uterine Artery Embolization for Uterine Fibroids
Brief Title: The FIRSTT: Comparing MRgFUS(MR-guided Focused Ultrasound) Versus UAE (Uterine Artery Embolization)for Uterine Fibroids.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Elizabeth A. Stewart, Professor of Obstetrics and Gynecology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-005095; 1RC1HD063312-01 (NIH)
Record Dates: First submitted 2009-10-13; First posted 2009-10-15 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Symptomatic Uterine Leiomyomas; Fibroids; Uterine Fibroids; Myomas
Keywords: Uterine fibroids; Fibroids; Uterine leiomyomas; UAE; UFE; Magnetic resonance guided focused ultrasound; MRgFUS; Pelvic pain
MeSH Terms: conditions — Leiomyoma; Myoma; Myofibroma; Pelvic Pain | interventions — Uterine Artery Embolization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Focused Ultrasound (MRgFUS) (Active Comparator)
  Interventions: Procedure: Focused ultrasound (MRgFUS)
- Uterine Artery Embolization (UAE) (Active Comparator)
  Interventions: Procedure: Uterine artery embolization (UAE)

INTERVENTIONS:
Procedure: Focused ultrasound (MRgFUS) — MRgFUS treatment will take place in a MRI machine and powerful ultrasound waves go through the abdominal wall to destroy the fibroid or fibroids. No incision is made during this treatment and light sedation is required. There are certain fibroids that may not be treated with this technique and there is no treatment of normal uterine tissue.ough the abdominal wall to destroy the fibroid.
  Other Names: ExAblate 2000
  Arms: Focused Ultrasound (MRgFUS)
Procedure: Uterine artery embolization (UAE) — UAE treatment takes place on a regular x-ray machine. A small incision is made where the leg meets the trunk and a small tube is used to use very small pellets to block off the blood supply to the entire uterus. Sedation is used. Most fibroids are treated with this technique and normal uterine tissue is also affected.
  Other Names: Uterine Fibroid Embolization; UFE
  Arms: Uterine Artery Embolization (UAE)

SUMMARY:
The primary goal of this study is to compare the safety and effectiveness of two standard fibroid treatments: MRI guided ultrasound surgery (MRgFUS) and uterine artery embolization (UAE). Both treatments are approved by the Food and Drug Administration (FDA) for women who do not plan to become pregnant.

A second goal of this study is to better understand which symptoms bother women with fibroids the most. Understanding and addressing the symptoms of clinically-significant uterine fibroids is important in order to optimize treatment outcomes and control health care costs.

Women who are eligible to participate in the study, are randomized to one of two treatment arms (UAE or MRgFUS). Women in both arms will receive treatment but will not be able to choose which treatment she will receive.

A comprehensive assessment of symptoms-including experienced pain- will take place at baseline, 6 weeks, and at 6, 12, 24, and 36 months following treatment with UAE and MRgFUS.

DETAILED DESCRIPTION:
Uterine fibroids affect up to 70 to 80% of women and about 30% of women are symptomatic. Over 200,000 hysterectomies are performed each year for uterine fibroids in the USA. The direct health care costs attributable to uterine fibroids exceed $2.1 billion annually. Fibroids are reported to cause a number of symptoms including heavy or prolonged menstrual bleeding, pelvic pressure, pain with menses and bowel and bladder dysfunction. However, fibroid symptomatology is incompletely understood. Understanding and addressing the myomas pain are important in optimizing treatment outcomes and controlling health care costs from a societal perspective. This study proposes to optimally characterize symptoms and symptom relief in women with leiomyomas severe enough to seek interventional therapy. Secondly we will characterize a variety of symptoms utilizing standardized instruments for other pelvic diseases and symptoms to optimize comparisons with other disease processes.

Clinical and scientific significance of the studies is high. We look to generate resources which can be used at a later time to assess the biologic and genetic variables affecting treatment outcome and to comprehensively assess the societal economic impact of uterine fibroids and their treatment with UAE and MRgFUS.

Participants will be in the study for up to 36 months following fibroid treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Women able to give informed consent and willing and able to attend all study visits
2. Premenopausal women at least 25 years of age
3. No evidence of High Grade SIL by pap smears or HPV testing within institutional guidelines.

Exclusion Criteria:

1. Women actively trying for pregnancy or currently pregnant
2. Uterine size > 20 weeks
3. Prior myomectomy, UAE, or MRgFUS. Previous hysteroscopic or laparoscopic myomectomy for the removal of only pedunculated leiomyomas (as described in #17, below) will be allowed and evaluated on an individual basis to determine eligibility for treatment.
4. More than 6 fibroids > than 3 centimeters in maximal diameter
5. Allergy to either gadolinium or iodinated contrast
6. Implanted metallic device prohibiting MRI
7. Severe claustrophobia
8. BMI which prohibits subject from fitting in MRI device
9. Severe abdominal scarring precluding safe MRgFUS treatment
10. Active pelvic infection
11. Intrauterine contraceptive device in place at the time of treatment
12. Current use of GnRH agonists or antagonists
13. Unstable medical conditions requiring additional monitoring during the procedure
14. Bleeding diathesis requiring medical treatment
15. Imaging suggestive of malignant disease of uterus, ovary, or cervix
16. Imaging suggestive of only adenomyosis
17. Pedunculated submucosal or subserosal myoma with a stalk less than 25% of the maximal fibroid diameter

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-04-29 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Symptomatic outcomes measured by validated instruments | At baseline, 6 weeks and 6, 12, 24, and 36 months following treatment.

SECONDARY OUTCOMES:
Adverse events following treatment | At baseline, 6 weeks and 6, 12, 24 and 36 months following treatment.
Biologic predictors of outcome | Blood sample is obtained at baseline and at 12, 24, and 36 months following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Stewart, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Health System, Durham, North Carolina

REFERENCES:
- [Derived] Laughlin-Tommaso SK, Gorny KR, Hesley GK, Vaughan LE, Woodrum DA, Lemens MA, Stewart EA. Uterine and Fibroid Imaging Analysis from the FIRSTT Study. J Womens Health (Larchmt). 2022 Apr;31(4):546-554. doi: 10.1089/jwh.2020.8892. Epub 2021 Jul 8. PMID 34242085
- [Derived] Laughlin-Tommaso S, Barnard EP, AbdElmagied AM, Vaughan LE, Weaver AL, Hesley GK, Woodrum DA, Jacoby VL, Kohi MP, Price TM, Nieves A, Miller MJ, Borah BJ, Moriarty JP, Gorny KR, Leppert PC, Severson AL, Lemens MA, Stewart EA. FIRSTT study: randomized controlled trial of uterine artery embolization vs focused ultrasound surgery. Am J Obstet Gynecol. 2019 Feb;220(2):174.e1-174.e13. doi: 10.1016/j.ajog.2018.10.032. Epub 2018 Oct 26. PMID 30696556
- [Derived] Barnard EP, AbdElmagied AM, Vaughan LE, Weaver AL, Laughlin-Tommaso SK, Hesley GK, Woodrum DA, Jacoby VL, Kohi MP, Price TM, Nieves A, Miller MJ, Borah BJ, Gorny KR, Leppert PC, Peterson LG, Stewart EA. Periprocedural outcomes comparing fibroid embolization and focused ultrasound: a randomized controlled trial and comprehensive cohort analysis. Am J Obstet Gynecol. 2017 May;216(5):500.e1-500.e11. doi: 10.1016/j.ajog.2016.12.177. Epub 2017 Jan 5. PMID 28063909
- [Derived] AbdElmagied AM, Vaughan LE, Weaver AL, Laughlin-Tommaso SK, Hesley GK, Woodrum DA, Jacoby VL, Kohi MP, Price TM, Nieves A, Miller MJ, Borah BJ, Gorny KR, Leppert PC, Lemens MA, Stewart EA. Fibroid interventions: reducing symptoms today and tomorrow: extending generalizability by using a comprehensive cohort design with a randomized controlled trial. Am J Obstet Gynecol. 2016 Sep;215(3):338.e1-338.e18. doi: 10.1016/j.ajog.2016.04.001. Epub 2016 Apr 9. PMID 27073063
- [Derived] Laughlin-Tommaso SK, Borah BJ, Stewart EA. Effect of menses on standardized assessment of sexual dysfunction among women with uterine fibroids: a cohort study. Fertil Steril. 2015 Aug;104(2):435-9. doi: 10.1016/j.fertnstert.2015.04.029. Epub 2015 May 16. PMID 25989973
- [Derived] Bouwsma EV, Hesley GK, Woodrum DA, Weaver AL, Leppert PC, Peterson LG, Stewart EA. Comparing focused ultrasound and uterine artery embolization for uterine fibroids-rationale and design of the Fibroid Interventions: reducing symptoms today and tomorrow (FIRSTT) trial. Fertil Steril. 2011 Sep;96(3):704-10. doi: 10.1016/j.fertnstert.2011.06.062. Epub 2011 Jul 27. PMID 21794858
- See also: National Institute of Child Health and Human Development — http://www.nichd.nih.gov/
- See also: Mayo Clinic Uterine Fibroids Information — http://www.mayoclinic.com/health/uterine-fibroids/DS00078
- See also: Radiology Society of North America Information on UFE — http://www.radiologyinfo.org/en/info.cfm?pg=ufe
- See also: Mayo Clinic Uterine Fibroid Facebook page sharing educational information related to fibroids. — http://on.fb.me/gewuoO